CLINICAL TRIAL: NCT00807001
Title: A Phase I/II, Double-Blind, Dose-Escalation Study to Evaluate the Safety and Antiviral Activity of IDX184 in Treatment-Naïve Subjects Infected With Genotype 1 Chronic Hepatitis C
Brief Title: Double-Blind, Dose-Escalation Study of IDX184 in Chronic Hepatitis C Treatment-Naïve Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2355-003; IDX-08C-003
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis C (HCV)
Keywords: Hepatitis C, HCV, treatment-naive
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — IDX184

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A (Experimental): Subjects randomized 8:2 (active:placebo) to receive one 25 milligrams (mg) capsule of IDX184 per day for 3 days. Fourteen days after treatment, subjects were offered a course of pegylated interferon and ribavirin according to local standard of care.
  Interventions: Drug: IDX184
- Cohort B (Experimental): Subjects randomized 8:2 (active:placebo) to receive two 25 mg capsules of IDX184 per day for 3 days. Fourteen days after treatment, subjects were offered a course of pegylated interferon and ribavirin according to local standard of care.
  Interventions: Drug: IDX184
- Cohort C (Experimental): Subjects randomized 8:2 (active:placebo) to receive three 25 mg capsules of IDX184 per day for 3 days. Fourteen days after treatment, subjects were offered a course of pegylated interferon and ribavirin according to local standard of care.
  Interventions: Drug: IDX184
- Cohort D (Experimental): Subjects randomized 8:2 (active:placebo) to receive four 25 mg capsules of IDX184 per day for 3 days. Fourteen days after treatment, subjects were offered a course of pegylated interferon and ribavirin according to local standard of care.
  Interventions: Drug: IDX184

INTERVENTIONS:
Drug: IDX184 — oral dose, active or placebo

SUMMARY:
This is a proof-of-concept study which will provide data about the safety and antiviral activity of several doses of the investigational drug IDX184 given for 3 days in treatment-naive HCV genotype 1-infected subjects so that optimal doses can be chosen for testing in later studies.

ELIGIBILITY:
Inclusion criteria:

1. 18-65 years old
2. Subject of childbearing potential must agree to use a consistent form of an acceptable double-barrier method of birth control.
3. Plasma HCV RNA ≥ 5 log10 IU/mL
4. HCV genotype 1

Exclusion criteria:

1. Received prior antiviral treatment for hepatitis C infection
2. Subject is pregnant or breastfeeding
3. Body Mass Index (BMI) > 32
4. Currently abusing alcohol or illicit drugs
5. Currently receiving methadone, buprenorphine or other drugs for the treatment of opioid addiction
6. Co-infected with hepatitis B virus (HBV, HBsAg positive) and/or human immunodeficiency virus (HIV)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

REFERENCES:
- [Result] Lalezari J, Asmuth D, Casiro A, Vargas H, Lawrence S, Dubuc-Patrick G, Chen J, McCarville J, Pietropaolo K, Zhou XJ, Sullivan-Bolyai J, Mayers D. Short-term monotherapy with IDX184, a liver-targeted nucleotide polymerase inhibitor, in patients with chronic hepatitis C virus infection. Antimicrob Agents Chemother. 2012 Dec;56(12):6372-8. doi: 10.1128/AAC.01521-12. Epub 2012 Oct 15. PMID 23070151

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | IDX184 25 mg | IDX184 50 mg | IDX184 75 mg | IDX184 100 mg
Started | 8 (For all groups, number of subjects who received at least one dose of study drug.) | 8 | 8 | 8 | 9
Completed | 8 | 7 | 8 | 8 | 9
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | IDX184 25 mg | IDX184 50 mg | IDX184 75 mg | IDX184 100 mg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 9 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (7.63) | 48.3 (6.50) | 48.8 (5.85) | 47.3 (8.12) | 47.2 (7.89) | 48.1 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 2 | 4 | 12
  Male | 5 | 6 | 7 | 6 | 5 | 29
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 8 | 7 | 7 | 36
  Argentina | 1 | 0 | 0 | 0 | 2 | 3
  Austria | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Adverse Event (Side Effect) and the Severity of Those Adverse Events
Description: Monitoring of adverse events, physical examination, routine safety laboratory parameters and electrocardiograms. 1=mild, 2=moderate, 3=severe, 4=potentially life-threatening
Time Frame: 17 days
Population: Safety population consisted of all subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | IDX184 25 mg | IDX184 50 mg | IDX184 75 mg | IDX184 100 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9
participants
  Number of subjects with any adverse event | 5 | 2 | 3 | 3 | 5
  Number of sub. with any Grade 3/4 lab abnormality | 1 | 1 | 0 | 0 | 2
  Grade 3/4 Triacylglycerol Lipase, high | 0 | 1 | 0 | 0 | 1
  Grade 3/4 Prothrombin Intl. Normalized Ratio, high | 0 | 0 | 0 | 0 | 1
  Grade 3/4 Prothrombin Time, high | 0 | 0 | 0 | 0 | 1
  Grade 3/4 Urine Erythrocytes, high | 0 | 0 | 0 | 0 | 1
  Grade 3/4 Pancreatic Amylase, high | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Antiviral Activity at Day 4. Change in Plasma HCV RNA (Hepatitis C Virus Ribonucleic Acid)
Description: Measures how much virus is in the blood.
Time Frame: Baseline to 4 days
Population: efficacy evaluable population = a) must have received all 3 doses of study drug b) must have baseline and at least one post-baseline HCV RNA determination
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Placebo | IDX184 25 mg | IDX184 50 mg | IDX184 75 mg | IDX184 100 mg
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 9
log10 IU/mL | -0.1 (0.3) | -0.5 (0.6) | -0.7 (0.2) | -0.6 (0.3) | -0.7 (0.5)

ADVERSE EVENTS:
Time Frame: 17 days
Arm/Group | Placebo | IDX184 25 mg | IDX184 50 mg | IDX184 75 mg | IDX184 100 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 5/8 | 2/8 | 3/8 | 3/8 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | IDX184 25 mg (N=8) | IDX184 50 mg (N=8) | IDX184 75 mg (N=8) | IDX184 100 mg (N=9)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Urinary sediment present (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Menopause (Social circumstances) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Adverse events summarized the 3 days of IDX184 dosing and 14 days of treatment free follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI that permits the sponsor to review results communications prior to public release and embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor may request the PI to remove the sponsor's confidential information prior to such publication.